CLINICAL TRIAL: NCT07216404
Title: Exploring the Safety, Acceptability, and Efficacy of Psilocybin Among Non-Small Cell Lung Cancer Patients With Major Depressive Disorder: A Proof-of-Concept Trial (DREAM LUNG STUDY)
Brief Title: Psilocybin-Assisted Therapy for the Treatment of Major Depressive Disorder in Patients With Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alan Davis (Other)
Responsible Party: Sponsor-Investigator, Alan Davis, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-24170; NCI-2025-06353 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-09-29; First posted 2025-10-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lung Non-Small Cell Carcinoma; Unipolar Depression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Depressive Disorder | interventions — Specimen Handling; Counseling; Interviews as Topic; Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (counseling sessions, psilocybin) (Experimental): Patients participate in two preparation therapy sessions over 4 hours each on days 7 and 14, then patients receive psilocybin PO on day 21 and participate in a single dosing therapy session for over 8-10 hours on study. Patients also complete two post-dosing therapy sessions over 2 hours each on days 22 and 28 on study. Patients additionally undergo blood and urine sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Counseling; Other: Interview; Drug: Psilocybin; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Counseling — Participate in therapy sessions
  Other Names: Counseling Intervention
Other: Interview — Ancillary studies
Drug: Psilocybin — Given PO
  Other Names: [3-[2-(dimethylamino)ethyl]-1H-indol-4-yl] dihydrogen phosphate
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase II trial tests the safety and side effects of psilocybin in combination with therapy for the treatment of major depressive disorder in patients with non-small cell lung cancer. A cancer diagnosis is life-changing, resulting in significant levels of psychological symptoms, including a combination of depression, anxiety, stress, including feelings of existential distress (i.e., loss of meaning, demoralization, despair). Among all cancer patients, those diagnosed with lung cancer have the highest prevalence of mood disorders, such as depression (up to 40%) leading to profound deterioration in quality of life, prolonged hospital stays, poorer treatment adherence, decreased survival rates, and high rates of suicide (5- and 3-times higher than the general population and other cancer patients, respectively). Psilocybin is substance being studied in the treatment of anxiety or depression in patients with advanced cancer. It is taken from the mushroom Psilocybe mexicana. Psilocybin acts on the brain to cause hallucinations (sights, sounds, smells, tastes, or touches that a person believes to be real but are not real). Psilocybin in combination with therapy may be safe and effective in treating major depressive disorder in patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and acceptability of psilocybin-assisted psychotherapy with non-small cell lung cancer (NSCLC) patients.

SECONDARY OBJECTIVE:

I. To determine the efficacy of psilocybin-assisted therapy in the reduction of depression and the impact of treatment on quality of life, cancer-related stress, and existential distress.

OUTLINE:

Patients participate in two preparation therapy sessions over 4 hours each on days 7 and 14, then patients receive psilocybin orally (PO) on day 21 and participate in a single dosing therapy session for over 8-10 hours on study. Patients also complete two post-dosing therapy sessions over 2 hours each on days 22 and 28 on study. Patients additionally undergo blood and urine sample collection throughout the study.

After completion of study treatment, patients are followed up at 4 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with NSCLC, confirmed by pathology report
* Have a Karnofsky performance status >= 60
* Participants receiving chemotherapy, radiation therapy, and biologic therapies may participate while receiving those therapies if they are tolerating the therapy or treatment sufficiently to allow administration of oral psilocybin and if treatments do not result in meeting any of the medical exclusion criteria outlined below
* Moderate to severe symptoms of depression (GRID Hamilton Rating Scale for Depression [GRID-HAMD] > 16)
* English-speaking
* Over the age of 18
* Have given written informed consent
* Able to read
* Be judged by study team clinicians to be at low risk for suicidality, as defined by a score of =< 2 on the Columbia- Suicide Severity rating scale (C-SSRS) ideation subscale, 0 on the behavior subscale, and by overall clinical judgment; and
* Have limited lifetime use of hallucinogens (the following criteria are preferred: no use in the past 5 years; total hallucinogen use less than 10 times)

Exclusion Criteria:

* GENERAL MEDICAL EXCLUSION CRITERIA
* Participants who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; participants who are of child-bearing potential and sexually active who are not practicing a highly effective means of birth control (i.e., implants, injectables, combined oral contraceptives, progestin containing intrauterine devices [IUDs], or vasectomized partner)
* Participants with partners of child-bearing potential who are sexually active and not practicing a highly effective means of contraception (i.e., condom with spermicidal foam/gel/film/cream/suppository)
* Cardiovascular conditions: Recent history of coronary artery disease or stroke, current uncontrolled angina, uncontrolled hypertension, a clinically significant electrocardiogram (ECG) abnormality as determined by a cardiologist and/or medical monitor (e.g., atrial fibrillation), prolonged corrected QT (QTc) interval (i.e., QTc > 450 msec), artificial heart valve, or transient ischemic attack (TIA) in the past year
* Systolic blood pressure (SBP) > 139 mm HG; diastolic blood pressure (DBP) > 89 mm HG; heart rate (HR) > 90 bpm (mean values of the four or more assessments will not exceed 139 mm Hg systolic, 89 mm Hg diastolic, and/or 90 beats per minute)
* Insulin-dependent diabetes
* Non-insulin dependent diabetes if recent history of symptomatic hypoglycemia
* Significant central nervous system (CNS) pathology. Some examples include:

  * Unstable primary or secondary (e.g., metastatic) cerebral neoplasm. Stable is defined as treatment within prior 4 weeks or no immediate plans for treatment.
  * Unstable history of seizures
  * Cerebral aneurysm - unstable with plans for intervention or close monitoring
  * Clinical diagnosis of dementia
  * Clinical diagnosis of delirium
* In the investigator's opinion, abnormal and clinically significant results on the physical examination, vital signs, ECG, or laboratory tests at screening may constitute a risk for an individual exposed to psilocybin. This includes platelets below 100,000 platelets per cubic millimeter of blood, liver function tests three times the upper limit of normal, and creatine two times above the normal range. This also includes clinically significant abnormal electrolytes or low hemoglobin (below 10 g/L)
* Any acute condition that would, in the Investigator's judgment, place the subject at significant risk due to safety concerns or compliance with clinical study procedures (e.g., electrolyte imbalance, infection/inflammation, intestinal obstruction, inability to swallow medication, etc.)
* Under active treatment of an investigational agent in a clinical trial
* In the judgement of the clinician, patients currently taking psychoactive medication on a regular (e.g., daily) basis (e.g., cannabis, opiates, Ritalin), other than a daily selective serotonin reuptake inhibitors (SSRI), serotonin-norepinephrine reuptake inhibitors (SNRI), or bupropion (< 300 mg daily) (Patients will not be instructed to hold prescribed psychoactive medications)
* In the judgement of the clinician, patients who self-report or urine test positive for psychoactive medications (e.g., illicit opiates, amphetamines, cocaine) may be excluded, for example recent use by self-report but urine test negative may still be enrolled, while participants with impaired mental status will be excluded
* PSYCHIATRIC EXCLUSION CRITERIA
* Current or past history of meeting Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or bipolar I or II disorder
* Current or history within one year of meeting DSM-5 criteria for a moderate or severe alcohol or other drug use disorder (excluding caffeine and tobacco)
* Have a first or second-degree relative with schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition) or bipolar I or II disorder
* Has a psychiatric condition that precludes the establishment of therapeutic rapport, as evidenced by long-term patterns of unstable relationships, a history of significant stress-related paranoia, and identity disturbances
* History of a medically significant suicide attempt as determined by the study team and principal investigator (PI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ratings of suicidal ideation on the Columbia- Suicide Severity rating scale (C-SSRS) | At baseline, one day post-drug session, and 4 weeks post-drug session
  Ratings of suicidal ideation on the C-SSRS will be summarized with means and standard deviations (SD) at baseline, one day post-drug session, and 4 weeks post-drug session. A mixed effects regression model will be fit containing a fixed effect for visit to test for a significant change in ratings of suicidal ideation from baseline to 4 weeks post drug session. Estimated mean differences will be presented with corresponding 95% confidence intervals (CI). An alpha level of 0.05 will be used to determine statistical significance.
Incidence of adverse events | At baseline, one day post-drug session, and 4 weeks post-drug session
  Descriptive analysis of adverse event reporting logs will be conducted to determine if any serious adverse events have been reported related to psilocybin administration.
Acceptability of psilocybin-assisted therapy | At end of visit 3 (7 days prior to drug administration) and 4 weeks post-drug session
  The mean (SD) change in Participant/Client Satisfaction Questionnaire levels between end of preparatory session 2 (visit 3; 7 days prior to drug administration) and 4 weeks post-drug session will be presented and a paired t-test will be used to test for a significant increase/decrease in acceptability. The estimated mean change will be presented with corresponding 95% confidence interval (CI). An alpha level of 0.05 will be used to determine statistical significance.
Satisfaction of psilocybin-assisted therapy | At end of visit 3 (7 days prior to drug administration) and 4 weeks post-drug session
  The mean (SD) change in Participant/Client Satisfaction Questionnaire levels between end of preparatory session 2 (visit 3; 7 days prior to drug administration) and 4 weeks post-drug session will be presented and a paired t-test will be used to test for a significant increase/decrease in satisfaction. The estimated mean change will be presented with corresponding 95% confidence interval (CI). An alpha level of 0.05 will be used to determine statistical significance.

SECONDARY OUTCOMES:
Depression symptom severity | At baseline, end of visit 3 (7 days prior to drug administration), and 4 weeks post-drug session.
  Mean (SD) ratings of depression symptom severity will be presented from baseline, end of preparatory session 2 (visit 3; 7 days prior to drug administration), and 4 weeks post-drug session. A mixed effects regression model will be fit containing a fixed effect for visit to test for a significant change in ratings of depressive symptom severity from baseline to 4 weeks post drug session. Estimated mean differences will be presented with corresponding 95% confidence intervals (CI). An alpha level of 0.05 will be used to determine statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Alan K Davis, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu